CLINICAL TRIAL: NCT03091491
Title: Randomised Phase 2 Study of Nivolumab Versus Nivolumab and Ipilimumab Combination in EGFR Mutant Non-small Cell Lung Cancer
Brief Title: Study of Nivolumab Verses Nivolumab and Ipilimumab Combination in EGFR Mutant Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment due to general pessimism for immunotherapy in NSCLC, availability of alternative therapy and clinician's choice to put patient on immunotherapy outside of trial setting.
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National University Hospital, Singapore (Other); Johns Hopkins Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-777
Record Dates: First submitted 2017-03-06; First posted 2017-03-27 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab (Experimental)
  Interventions: Drug: Nivolumab
- Nivolumab and Ipilimumab (Experimental)
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 1 mg/kg administered every 6 weeks as a 30 min IV infusion
  Other Names: Yervoy
  Arms: Nivolumab and Ipilimumab
Drug: Nivolumab — Nivolumab 3 mg/kg administered every 2 weeks as a 30 min IV infusion
  Other Names: Opdivo

SUMMARY:
The purpose of this study is to determine whether Nivolumab in combination with Ipilimumab is associated with superior response rate compared to Nivolumab alone in patients with advanced Epidermal Growth Factor Receptor (EGFR) mutation positive Non-small Cell Lung Cancer who have failed one line of standard EGFR tyrosine kinase inhibitor and not more than one line of chemotherapy regimen. This study also aims to determine predictive biomarkers of response/benefit in patients with EGFR mutation positive NSCLC.

DETAILED DESCRIPTION:
This study examines the outcome of nivolumab single agent versus nivolumab-ipilimumab combination in patients with advanced EGFR+ NSCLC who have failed one line of standard EGFR Tyrosine Kinase Inhibitor (TKI) and not more than one line of chemotherapy regimen. The use of 3rd generation EGFR TKI for patients with acquired mutation that substitute a threonine (T) with a methionine (M) at position 790 of exon 20 (T790M) is allowed.

Patients will be randomized in a 1:1 ratio to treatment with either nivolumab monotherapy (Arm A) or nivolumab/ipilimumab combination therapy (Arm B) and will be stratified according to the following factors:

* Programmed Death-Ligand 1 (PDL1) status: <1% vs ≥1%
* Presence of brain metastasis
* Institution: National Cancer Centre Singapore, National University Cancer Institute, and Johns Hopkins Singapore-Tan Tock Seng Hospital

Both arms will continue with treatment regimen till disease progression or discontinuation of treatment due to adverse events.

Arm A patients are allowed to cross over to Arm B in the event of clear-cut disease progression.

On-study tumor assessments will be conducted every 6 weeks for 24 weeks and then every 12 weeks till clear-cut disease progression.

The radiologist will be blinded to the treatment arm that the patient is randomised to ensure an objective response evaluation.

ELIGIBILITY:
Inclusion Criteria:

i. Signed informed consent

ii. Male or female, 21 years or older

* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 5 months (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab
* Women must not be breastfeeding
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception
* WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 milli-international units per millilitre (mIU/mL).
* Women of childbearing potential (WOCBP) receiving nivolumab will be instructed to adhere to contraception for a period of 5 months after the last dose of investigational product. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. These durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days and men who are sexually active with WOCBP use contraception for 5 half-lives plus 90 days.

iii. Advanced EGFR+ NSCLC

iv. Eastern Cooperative Oncology Group (ECOG) 0-2 performance status

v. Progressed on one line of standard EGFR TKI and not more than one line of chemotherapy; 3rd generation EGFR TKI for patients with T790M mutation is allowed

* A 14-day washout period is required for EGFR TKI for patients who received this as the last therapy before recruitment
* A 28-day washout period is required for chemotherapy for patients who received this as the last therapy before recruitment. All drug-related toxicities should have returned to baseline with the exception of neuropathy, fatigue, and alopecia.

vi. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to randomization/registration

* White Blood Cell (WBC) ≥ 2000/µL
* Neutrophils ≥ 1000/µL
* Platelets ≥ 100 x 10^3/µL
* Hemoglobin > 9.0 g/dL
* Serum creatinine ≤ 1.5 x Upper Limit of Normal (ULN) or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula below):
* Aspartate Aminotransferase/ Alanine Aminotransferase (AST/ALT) ≤ 3 x ULN
* Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)

vii. Measurable disease, as defined by RECIST v1.1; Previously irradiated lesions can only be considered as measurable disease if disease progression has been unequivocally documented at that site since radiation.

viii. Patients with a history of treated asymptomatic central nervous system (CNS) metastases are eligible, provided they meet all of the following criteria:

1. Measurable disease outside CNS
2. No ongoing requirement for corticosteroids as therapy for CNS disease; anticonvulsants at a stable dose allowed
3. No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to randomization
4. No evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study

ix. Tumor sites amenable for CT-guided core biopsies or trucut biopsies

x. Willing to undergo 2 biopsies and contribute research bloods for the study. Archived tissue that is less than 6 months old is acceptable as an alternative to biopsy at screening if a biopsy is not feasible; patients from arm A must be willing to undergo biopsy as baseline upon clear-cut disease progression and on-treatment repeat biopsy before they are allowed to cross over to receive ipilimumab in addition to nivolumab.

xi. Patients with confirmed concomitant HBV infection that are eligible for inclusion must be treated with antiviral therapy prior to enrollment to ensure adequate viral suppression (HBV DNA < 2000 IU/mL), must remain on antiviral therapy for the study duration, and continue therapy for 6 months after the last dose of investigational product(s). Subjects with confirmed Hepatitis C (HCV) infection who are negative for HBsAg and positive for anti-HBc, are eligible but must be started on active antiviral therapy (for HBV) prior to their first dose of investigational product.

xi. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception and to continue its use for 90 days after the last dose of nivolumab

xii. Women who are not postmenopausal (≥12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 24 hours prior to initiation of study drug

xiii. Available for follow-up

Exclusion Criteria:

i. Symptomatic brain or leptomeningeal metastases (patients who have treated stable brain or Leptomeningeal disease are eligible; there is no magnetic resonance imaging (MRI) evidence of progression for [lowest minimum is 4 weeks or more] after treatment is complete and within 28 days prior to the first dose of nivolumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration).

ii. Poor performance status of ECOG 3-4

iii. Tumour sites not amenable to CT-guided core biopsies or trucut biopsies; However waiver for this criterion can be given for selected patients on a case-by-case basis for patients with sites of disease that are technically difficult to access after discussion with interventional radiologist. Waivers are allowed for not more than 70 patients for this study in order to allow sufficient number of quality tumour biopsies for biomarker analysis in this study. Waivers would have to be approved by the Principal Investigator.

iv. Unwilling to undergo 2 biopsies and contribute research bloods for the study

v. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins

vi. Concurrent Autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.

vii. Prior treatment with other anti-Programmed cell death protein 1 (anti-PD1) or anti-PDL1 or anti-CTLA4 therapies

viii. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (anti-TNF) agents) within 2 weeks prior to randomization

1. Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study.
2. Patients with history of allergic reaction to IV contrast requiring steroid pre-treatment should have baseline and subsequent tumor assessments done by MRI.
3. The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.

ix. Active interstitial lung disease or history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan; History of radiation pneumonitis in the radiation field (fibrosis) is permitted.

x. Active tuberculosis

xi. Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)

xii. Prior allogeneic bone marrow transplantation or solid organ transplant

xiii. Administration of a live, attenuated vaccine within 4 weeks before randomization or anticipation that such a live attenuated vaccine will be required during the study

xiv. Not available for follow-up and unlikely to be compliant with follow-up or protocol requirements

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | From baseline until best overall response of Complete Response (CR) or Partial Response (PR), up to 2 years

SECONDARY OUTCOMES:
Progression-Free Survival | From time of randomisation until first documented disease progression or death due to any cause, up to 2 years
Duration of Response | From time of first response until first documented disease progression or death due to any cause, up to 2 years
Overall Survival | From time of randomisation until death due to any cause, up to 2 years
Evaluate the toxicity profiles of Nivolumab with or without Ipilimumab by measuring the number of participants with treatment-related adverse events | From the time the Informed Consent Form is signed until at least 100 days after discontinuation of dosing, up to 2 years
  Safety data of all adverse events and serious adverse events, will be graded according to the NCI CTCAE v 4.0.
Evaluate capability of the addition of Ipilimumab to patients who progress on Nivolumab alone (Arm A) to achieve clinical benefit by measuring the time taken to achieve CR, PR or Stable Disease (SD) | From time of first dose of Ipilimumab until best overall response of CR, PR, or SD, up to 2 years
Evaluate an array of biomarkers in predicting response to Nivolumab and/or Ipilimumab | From time of first dose of study treatment until clear-cut disease progression, up to 2 years
  Biomarkers: PD-L1, mutational burden, microsatellite instability, blood-based biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Eng Huat Tan, Principal Investigator — National Cancer Centre, Singapore
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided